CLINICAL TRIAL: NCT04975373
Title: Reduction of Intrauterine Adhesions by Intrauterine Hyaluronic Acid Gel After Hysteroscopic Removal of Retained Products of Conception: Multicenter Prospective Randomized Trial
Brief Title: Intrauterine Hyaluronic Acid Gel for Prevention of Intrauterine Adhesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Barzilai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0002-21
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Prevenetion of Intrauterine Adhesions by Hyaluronic Acid Gel
Keywords: retained placenta; operative hysteroscopy; intrauterine adhesions; hyaluronic acid
MeSH Terms: conditions — Placenta, Retained; Gynatresia | interventions — Hysteroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Other): study group women in this group will receive intrauterine hyaluronic acid injection after operative hysteroscopy
  Interventions: Drug: Intrauterine injection of hyaluronic acid
- control group (No Intervention): women will not receive hyaluronic acid after operative hysteroscopy

INTERVENTIONS:
Drug: Intrauterine injection of hyaluronic acid — operative hysteroscopy - as a part of treatment in cases with retained placenta after delivery diagnostic hysteroscopy - as a routine evaluation after removal of placenta
  Other Names: operative hysteroscopy -; diagnostic hysteroscopy
  Arms: study group

SUMMARY:
Women undergoing operative hysteroscopy for removal of retained placenta after delivery will be randomized into two groups.

1. study group - immediately after operative hysteroscopy 5 ml hyaluronic acid gel will be injected into uterine cavity
2. control group - no injection

4-8 weeks after operative hysteroscopy, participants will undergo diagnostic hysteroscopy with no anesthesia , as a part of routine evaluation after removal of retained placenta in Israel.

during diagnostic hysteroscopy the uterine cavity will be evaluated and the presence of adhesions and severity of adhesions will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing hysteroscopic removal of retained placenta after delivery

Exclusion Criteria:

* Known adverse reaction or allergy to hyaluronic acid

History of intrauterine adhesions

Acute pelvic inflammatory disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-07-25 (Estimated); Study Completion 2022-07-25 (Estimated)

PRIMARY OUTCOMES:
any adhesions | 4-8 weeks after intervention
  presence of any adhesions in uterine cavity during diagnostic hysteroscopy

SECONDARY OUTCOMES:
adhesion scorring | 4-8 weeks after intervention
  American Fertility Society score for intrauterine adhesions

CONTACTS AND LOCATIONS:
Locations (1):
- Barzilai University Medical Center, Ashkelon, Israel

IPD SHARING:
Plan to Share IPD: No